CLINICAL TRIAL: NCT07375641
Title: The Effect of Age and Sex on Pre-procedural Anticipated Pain and Post-procedural Experienced Pain in Patients Undergoing Flexible Cystoscopy for the First Time in an Outpatient Setting
Brief Title: The Impact of Age and Sex on Anticipated and Experienced Pain in First-Time Outpatient Flexible Cystoscopy
Acronym: PAINCYST
Status: Not yet recruiting | Type: Observational
Sponsor: Kayseri Education and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Abdullah Gölbaşi, Assitant Professor Abdullah Gölbaşı, Kayseri Education and Research Hospital
Other Study IDs: SBU-URO-AG-03
Record Dates: First submitted 2026-01-22; First posted 2026-01-29 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Urethral Stricture; Bladder (Urothelial, Transitional Cell) Cancer; Benign Prostate Obstruction (BPO)
Keywords: flexible cystoscopy; outpatient urology; pain perception
MeSH Terms: conditions — Urethral Stricture; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- First-Time Flexible Cystoscopy Under Local Anesthesia Patient Group: Patients who undergo flexible cystoscopy for the first time under local anesthesia in an outpatient clinic and are evaluated for pain

SUMMARY:
Cystoscopy is a procedure frequently performed in daily urological practice for the diagnosis of various urological conditions, including bladder tumors, benign prostatic hyperplasia, recurrent cystitis, and urethral strictures. Cystoscopy can be performed either in the operating room under sedation, spinal anesthesia, or general anesthesia, or in the outpatient setting under local anesthesia. Performing cystoscopy under outpatient conditions for patients requiring the procedure for follow-up and treatment indications is important in terms of reducing the workload of operating rooms. Although cystoscopy is generally well tolerated under local anesthesia in the outpatient setting, it may cause pain and anxiety in some patients, even when a flexible cystoscope is used. This may lead to adverse outcomes, particularly in patients with bladder tumors, due to loss to follow-up. Despite the use of analgesic methods such as lidocaine-based lubricants to reduce pain and anxiety before cystoscopy, an optimal solution has not yet been achieved. Moreover, some studies have reported that the level of pain experienced during cystoscopy increases with advancing age.

In male patients, several studies have demonstrated that the most painful moment during cystoscopy occurs when the tip of the cystoscope passes through the external urinary sphincter. It has been shown that asking patients to take deep breaths or allowing them to watch cystoscopy videos while manually compressing the irrigation fluid bag during the passage of the cystoscope through the bulbar urethra, just distal to the external urinary sphincter, can reduce pain perception. Female patients tend to experience less pain due to the shorter urethral length. Various strategies have been employed to minimize pain and anxiety during the procedure, including listening to music, watching relaxing videos, or allowing patients to view their own cystoscopy recordings during the examination. Given the lack of prior cystoscopy experience, we planned this randomized prospective study to evaluate the effect of age and sex on pain perception during flexible cystoscopy. We believe that the findings of this study may be beneficial in counseling patients during cystoscopic evaluation of urological pathologies

DETAILED DESCRIPTION:
Cystoscopy is one of the most commonly performed diagnostic procedures in daily urological practice and is widely used for the diagnosis and follow-up of various urological conditions, including bladder tumors, benign prostatic hyperplasia, recurrent lower urinary tract infections, evaluation of hematuria, and urethral strictures. Owing to its ability to allow direct visualization of the urothelial surface, cystoscopy provides high diagnostic accuracy and serves as a valuable tool in guiding treatment planning.

Depending on the patient's clinical status, comorbidities, and the indication for the procedure, cystoscopy may be performed in the operating room under sedation, spinal anesthesia, or general anesthesia, or safely conducted in the outpatient setting under local anesthesia. Performing cystoscopy in outpatient conditions, particularly for surveillance and follow-up purposes, is of considerable importance in terms of optimizing healthcare resources. Outpatient cystoscopy reduces operating room workload, eliminates anesthesia-related risks, shortens procedural time, and lowers overall healthcare costs.

Although the development of flexible cystoscopes has significantly improved patient comfort compared with rigid instruments, cystoscopy performed under local anesthesia in the outpatient setting may still cause substantial pain, discomfort, and anxiety in a subset of patients. This issue is of particular clinical relevance in patients with bladder tumors who require regular cystoscopic surveillance, as negative procedural experiences may result in poor compliance and loss to follow-up, potentially leading to delayed diagnosis and adverse oncological outcomes.

Various analgesic and anxiolytic strategies have been employed to alleviate pain and anxiety prior to cystoscopy, most commonly the use of lidocaine-based lubricating gels. In addition, adequate patient information, proper positioning, and gentle instrumentation are routinely applied to improve procedural tolerance. However, current evidence suggests that none of these approaches alone is sufficient to completely eliminate pain and anxiety, and an optimal, universally accepted strategy has yet to be established.

Several studies have reported that pain perception during cystoscopy may be influenced by patient age, with higher pain scores observed in older individuals. This association has been attributed to age-related changes in urethral and bladder neck elasticity, the presence of lower urinary tract symptoms, and increased comorbid conditions in elderly patients.

Sex-related differences also play a significant role in pain perception during cystoscopy. In male patients, previous studies have demonstrated that the most painful phase of the procedure occurs when the tip of the cystoscope passes through the external urinary sphincter. Increased resistance encountered during passage through the bulbar urethra, located immediately distal to the external sphincter, has been associated with heightened pain perception. It has been shown that simple manual compression of the irrigation fluid bag combined with instructing patients to take deep breaths or allowing them to watch cystoscopy videos during this phase can significantly reduce perceived pain.

In contrast, female patients generally report lower pain scores during cystoscopy, which is primarily attributed to the shorter length and more straightforward anatomical course of the female urethra, resulting in shorter procedural duration and less resistance during instrument insertion.

In recent years, increasing attention has been directed toward non-pharmacological interventions aimed at minimizing pain and anxiety during cystoscopy. Techniques such as listening to music, watching relaxing videos, or allowing patients to view their own cystoscopy recordings in real time have been shown to improve patient comfort and reduce pain perception during the procedure.

In light of these findings, we designed this randomized prospective study to evaluate the effect of age and sex on pain perception during flexible cystoscopy in male and female patients aged 18 years and older with no prior history of cystoscopy. We hypothesized that a better understanding of these factors would be beneficial for patient counseling and may improve patient compliance during cystoscopic evaluation of urological pathologies.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Patients undergoing flexible cystoscopy for the first time under local anesthesia in an outpatient setting
* Ability to understand the study procedures and provide informed consent

Exclusion Criteria:

* Use of systemic analgesics, sedatives, or anxiolytics immediately before the procedure
* Presence of active urinary tract infection at the time of cystoscopy
* Presence of an indwelling urethral catheter at the time of cystoscopy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients (≥18 years) undergoing first-time flexible cystoscopy under local anesthesia in an outpatient setting, with assessment of expected and perceived pain levels
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Correlation between expected pain and perceived pain | Immediately after completion of the cystoscopy procedure
  Correlation between pre-procedural expected pain scores and post-procedural perceived pain scores with using a validated pain scale of Visual Analog Scale [VAS]

SECONDARY OUTCOMES:
Pre-procedural expected pain level | Immediately before flexible cystoscopy
  Expected pain level assessed immediately before the procedure using a validated pain scale (e.g., Visual Analog Scale [VAS], 0-10)
Difference between expected and perceived pain levels | From immediately before to immediately after the procedure
  Difference between pre-procedural expected pain score and post-procedural perceived pain score
Effect of age on pain perception | Immediately after the procedure
  Association between patient age and post-procedural pain intensity during flexible cystoscopy
Effect of sex on pain perception | Immediately after the procedure
  Comparison of post-procedural pain intensity between male and female patients undergoing first-time flexible cystoscopy

CONTACTS AND LOCATIONS:
Overall Officials: Mert Karadağ, Professor, Study Chair — Kayseri Education and Research Hospital
Locations (1):
- Kayseri Education and Research Hospital, Kayseri, Kocasinan, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No